CLINICAL TRIAL: NCT04159662
Title: Brain Imaging of Cognition Inn Schizophrenia and Depression
Status: Recruiting | Type: Observational
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Synthia Guimond, Scientist, The Royal Ottawa Mental Health Centre
Other Study IDs: 2018037
Record Dates: First submitted 2019-10-25; First posted 2019-11-12 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia / Schizoaffective Disorder; Depression / Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with Schizophrenia or Schzioaffective Disorders: Clinical group
- Individuals with Major Depressive Disorder: Clinical group
- Healthy Individuals: Control group

SUMMARY:
Schizophrenia and depression are among the most disabling disorders in all of medicine. Cognitive deficits play a key role in patients' disability, affecting their capacity to contribute actively to society by sustaining employment or academic activity. Moreover, cognitive difficulties tend to persist even after the stabilization of other clinical symptoms. Verbal memory and emotion regulation are two important cognitive domains that are impaired in schizophrenia and depression and are associated with patients' functional outcomes. In this study, we are using brain imaging to investigate the brain mechanisms underlying these cognitive deficits in these populations.

DETAILED DESCRIPTION:
This study uses Functional Magnetic Resonance Imaging (fMRI) to help us better understand the cognitive problems that people who have schizophrenia, schizoaffective disorder, or depression experience. Cognitive problems can encompass a variety of different domains such as with attention, thinking, memory, emotion, and emotional regulation.

The study will involve three visits at The Royal's Institute of Mental Health Research. Each visit will last about 2.5 hours long.

Visits 1 and 2: We ask participants to fill out several questionnaires on a computer. We also ask participants to answer some questions about their current and past mental health. Participants will also perform some tasks involving general thinking skills.

Visit 3: This is the scan visit where we use fMRI, which is a technique that allows us to take a 3D picture of the brain using magnetic fields. It also allows us to estimate how active different regions of the brain are. During the fMRI, participants will lay down in a narrow tube in the fMRI scanner and hold still. Throughout the experiment, participant will perform three short tasks in the scanner, where they will see words and pictures and press a button to answer some questions.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* current Intelligence Quotient (IQ) > 70 as measured by the Wechsler Abbreviated Scale of Intelligence (WASI)
* the ability to read and speak fluent English
* a diagnosis of schizophrenia, schizoaffective or major depression disorder
* stable medication for more than one month

Exclusion Criteria:

* significant neurological or other medical disorders that may produce cognitive impairment
* a recent history of substance abuse or dependence (within the past 3 months)
* any magnetic resonance imaging (MRI) contraindications (e.g. metallic head implant, history of seizure, pacemaker)
* decisional incapacity requiring a guardian
* taking medications that are rated as Anticholinergic Burden (ACB) Score 3 (severe) or taking benzodiazepines on a daily basis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with an official diagnosis of: Schizophrenia, Schzioaffective or Major Depressive Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in verbal memory performance from baseline - Hopkins Verbal Learning Test-Revised (HVLT-R) | baseline, mid-treatment (3 weeks) and post treatment (7 weeks)
  The Hopkins Verbal Learning Test - Revisited (HVLT-R) for verbal memory is a 12-item test to measure a person's ability to encode, combine, store and recover verbal information in memory.
Change in emotion regulation performance from baseline - Mayer-Salovey-Caruso Emotional Intelligence Test (MSECIT) | baseline, mid-treatment (3 weeks) and post treatment (7 weeks)
  The Mayer-Salovey- Caruso Emotional Intelligence Test (MSCEIT) is a 141-item ability-based test designed to measure the four branches of emotional intelligence model of Mayer and Salovey (including emotion regulation).

SECONDARY OUTCOMES:
Change in composite scores on cognitive assessments from baseline | baseline and post treatment (7 weeks)
  Assessed with a battery of standardized tests examining cognitive capacity. These tests measure various cognitive domains such as attention, memory, executive function, speed of processing and emotion recognition.
Change in brain activity from baseline | baseline and post treatment (8 weeks)
  Brain activity as measured using resting-state and task-based functional magnetic resonance imaging (fMRI).

OTHER OUTCOMES:
Change in composite scores on social functioning from baseline | baseline and post treatment (9 weeks)
  Assessed with a battery of standardized tests examining social functioning. These tests measure an individual's level of social and occupational functioning as well as performance on everyday functional tasks (e.g., making phone calls, counting change, etc.).
Change in symptom severity from baseline - Positive and Negative Syndrome Scale (PANSS) | baseline and post treatment (9 weeks)
  The Positive and Negative Syndrome Scale (PANSS) is a 30-item medical scale used for measuring symptom severity of patients with schizophrenia. Total scores range from 30 to 210, with a larger score indicating greater severity of symptoms.
Change in perceived cognitive impairments from baseline - Subjective Scale to Investigate Cognition in Schizophrenia - Brief (SSTICS-B) | baseline and post treatment (9 weeks)
  The Subjective Scale to Investigate Cognition in Schizophrenia - Brief (SSTICS-B) is a self-rated 14-item scale that assesses the subjective level of cognitive abilities over the past week, ranging from "never" to "very often". The total score of SSTICS ranges from 0 to 84, with a greater score indicating greater perceived cognitive impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Synthia Guimond, PhD, Principal Investigator — Royal Ottawa Mental Health Centre
Locations (1):
- Royal Ottawa Mental Health Center, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected from this study may be shared with other researchers at the Royal's Institute of Mental Health Research for analyses and re-analyses. Variables of the study and scripts used for analyses will be made available to the public. De-identified data will also be shared with the general public upon request. Data that can connect with participants' identity will NOT be used or shared for analyses.
Supporting Information: SAP, Analytic Code
Time Frame: De-identified data will become available upon completion of the study and once results have been published in an academic journal (anticipated time frame: the year of 2024).